CLINICAL TRIAL: NCT00632840
Title: Regulation of Lipoprotein Kinetics by Atorvastatin and Fenofibrate With the Metabolic Syndrome
Brief Title: Pharmacological Regulation of Fat Transport in Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Western Australia (Other)
Collaborators: National Heart Foundation, Australia (Other)
Responsible Party: Gerald F Watts, University of Western Australia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UWA_DC012008
Record Dates: First submitted 2008-02-20; First posted 2008-03-11 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-02

CONDITIONS: Obesity; Lipid Disorders; Hypertriglyceridemia; Cardiovascular Disease
MeSH Terms: conditions — Obesity; Lipid Metabolism Disorders; Hypertriglyceridemia; Cardiovascular Diseases | interventions — Atorvastatin; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- P (Placebo Comparator): placebo group
  Interventions: Drug: Atorvastatin and fenofibrate
- Feno (Active Comparator): Fenofibrate
  Interventions: Drug: Atorvastatin and fenofibrate
- ATV (Active Comparator): Atorvastatin
  Interventions: Drug: Atorvastatin and fenofibrate

INTERVENTIONS:
Drug: Atorvastatin and fenofibrate — atorvastatin (40mg/day) fenofibrate (200mg/day)
  Other Names: Lipitor; Lofibra

SUMMARY:
The purpose of this study is to determine whether atorvastatin and fenofibrate are effective in the treatment of lipid disorders in obese, insulin resistant subjects.

DETAILED DESCRIPTION:
Insulin resistance is a heterogeneous metabolic disorder of complex etiology. It underpins dyslipoproteinemia, a key feature of the metabolic syndrome (MetS) that independently predicts cardiovascular disease (CVD). Hypertriglyceridemia, the most consistent lipid disorder in subjects with obesity and type 2 diabetes mellitus, is chiefly a consequence of overproduction and delayed clearance of triglyceride-rich lipoproteins (TRLs). Although the precise mechanisms involved are incompletely understood, experimental and clinical evidence suggests that elevated apolipoprotein (apo) C-III may play a crucial role in the dysregulation of TRL metabolism. investigating the effects of these agents on VLDL-apoC-III kinetics. In this study, we aimed to examine the effect of two lipid-regulating agents, atorvastatin and fenofibrate on VLDL-apoC-III transport. We hypothesized that atorvastatin and fenofibrate would have similar effects on apoC-III transport by decreasing the production and increasing the catabolism of VLDL-apoC-III.

ELIGIBILITY:
Inclusion Criteria:

any three of the followings

* waist circumference >102cm
* triglycerides >1.7 mmol/L
* HDL-cholesterol <1.05 mmol/L
* blood glucose >6.1 mmol/L
* blood pressure >130/85mmHg

Exclusion Criteria:

* plasma cholesterol >7mmo/L
* triglycerides >4.5mmo/L
* diabetes mellitus (defined by oral glucose tolerance test)
* CVD
* consumption of >30g alcohol/day
* use of agents affecting lipid metabolism
* APOE2/E2 genotype, macroproteinuria
* creatinaemia (>120umol/L)
* hypothyroidism
* abnormal liver and muscle enzymes.

Ages: 25 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2001-06; Primary Completion 2002-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
VLDL-apoC-III transport rate | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dick C Chan, PhD, Principal Investigator — The University of Western Australia

REFERENCES:
- [Derived] Chan DC, Watts GF, Ooi EM, Rye KA, Ji J, Johnson AG, Barrett PH. Regulatory effects of fenofibrate and atorvastatin on lipoprotein A-I and lipoprotein A-I:A-II kinetics in the metabolic syndrome. Diabetes Care. 2009 Nov;32(11):2111-3. doi: 10.2337/dc09-0519. Epub 2009 Aug 3. PMID 19651918
- [Derived] Chan DC, Barrett PH, Ooi EM, Ji J, Chan DT, Watts GF. Very low density lipoprotein metabolism and plasma adiponectin as predictors of high-density lipoprotein apolipoprotein A-I kinetics in obese and nonobese men. J Clin Endocrinol Metab. 2009 Mar;94(3):989-97. doi: 10.1210/jc.2008-1457. Epub 2008 Dec 30. PMID 19116237